CLINICAL TRIAL: NCT07052877
Title: Investigating Glioblastoma PSMA Expression by Utilizing Anti-VEGF and Its Effect on PSMA PET Scan Avidity
Brief Title: The Effect of Glioblastoma PSMA Expression Following Tumour VEGF Blockade From Bevacizumab
Acronym: GUAVA
Status: Not yet recruiting | Type: Observational
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Alexander Yuile, Principal Investigator, Royal North Shore Hospital
Other Study IDs: GUAVA
Record Dates: First submitted 2025-06-23; First posted 2025-07-07 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; Glioblastoma Multiforme (GBM)
Keywords: glioblastoma; anti-VEGF; PSMA; bevacizumab; VEGF; glioma; astrocytoma
MeSH Terms: conditions — Glioblastoma; Glioma; Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples including plasma.
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with glioblastoma receiving Bevacizumab as part of their standard of care
  Interventions: Diagnostic Test: PSMA PET/CT scan

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT scan — PSMA PET scan will be used to monitor changes in PSMA expression in response to bevacizumab.

SUMMARY:
This trial is a single arm study for patients receiving bevacizumab for IDH-wildtype glioblastoma. Patients receiving bevacizumab (an anti-VEGF therapy) will receive PSMA scans to investigate the role of PSMA expression in glioblastoma and its relationship to VEGF expression.

ELIGIBILITY:
Inclusion Criteria:

* > 18 year of age
* ECOG 0-2
* Able to provide informed consent for the study
* Minimum of 1 month from completion of radiotherapy with clinical or radiography evidence suggesting residual tumour
* Confirmed glioblastoma IDH1/2 wildtype (WHO2021)
* For bevacizumab treatment as per treating physician
* Able to comply with trial requirements

Exclusion Criteria:

* No major organ impairment that would likely lead to unacceptable toxicities- eg significant cardiac, hepatic, renal or haematologic dysfunction (based on clinician assessment)
* Any contraindication to bevacizumab, MRI gadolinium contrast or 68Ga-PSMA-617 radioisotope
* Any implant, foreign body, 3T MRI incompatible device or other contraindication to MRI imaging
* Does not fulfill PBS requirements for bevacizumab
* Women lactating, pregnant or of child baring potential who are not willing to avoid pregnancy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioblastoma patients receiving Bevacizumab as part of standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Changes in PSMA PET metabolic tumour volume (MTV) before and after bevacizumab administration. | Prior to first administration of bevacizumab to 6 weeks after.

OTHER OUTCOMES:
Changes in PSMA PET SUVmax before and after bevacizumab administration. | Prior to first administration of bevacizumab to 6 weeks after.
Changes in PSMA PET SUVmean before and after bevacizumab administration. | Prior to first administration of bevacizumab to 6 weeks after.
Changes in PSMA PET SUVpeak before and after bevacizumab administration. | Prior to first administration of bevacizumab to 6 weeks after.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal North Shore Hospital, Saint Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No